CLINICAL TRIAL: NCT02312765
Title: Reducing Heart Failure Re-admissions by Enhancing Sleep Apnea Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: AirCare Labs, LLC (Unknown)
Responsible Party: Principal Investigator, Nalaka Gooneratne, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 820241
Record Dates: First submitted 2014-12-01; First posted 2014-12-09 (Estimated); Results first posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Congestive Heart Failure; Sleep Apnea Syndromes
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Study participants will receive a tablet computer with the AirCare system.
  Interventions: Behavioral: AirCare App
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: AirCare App — Tablet software to encourage adherence and support
  Arms: Intervention

SUMMARY:
Sleep apnea, characterized by abnormal breathing at night, is often untreated in patients with heart failure. Helping patients to effectively use the most common form of treatment for sleep apnea, positive airway pressure therapy, can improve their heart function. This can reduce the likelihood that the patient will be re-admitted to the hospital. AirCareLabs has developed an innovative solution that allows patients to communicate with health care providers 24 hours a day, thus allowing them to get the help they need to effectively use positive airway pressure and thereby reduce the risk of being re-admitted to the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure and sleep apnea

Exclusion Criteria:

* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-11; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nalaka Gooneratne, MD, Study Director — University of Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: AirCare System: Study participants will receive a tablet computer with the AirCare system.
  AirCare App: Tablet software to encourage adherence and support
- Control: Standard of Care: Standard care consisting of routine clinical care provided by their healthcare providers
Period: Overall Study
Arm/Group | Intervention: AirCare System | Control: Standard of Care
Started | 74 | 72
Completed | 19 | 36
Not Completed | 55 | 36

BASELINE CHARACTERISTICS:
Population: Patients admitted with heart failure
Groups:
- Control: Standard of Care: Standard care: This is the care that would be routinely provided by their healthcare provider
- Total: Total of all reporting groups
Arm/Group | Intervention: AirCare System | Control: Standard of Care | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (11.9) | 59.4 (12.7) | 58.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 43 | 46 | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 43 | 33 | 76
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 19 | 30 | 49
Apnea Hypopnea Index (AHI, events/hr) [Mean (Standard Deviation); unit: events/hr] — The number of apnea (cessation of breathing) or hypopnea (reduction of breathing) events as defined by the American Academy of Sleep Medicine. Lowest possible value is 0 events per hour. Higher values indicate more frequent apnea or hypopnea events.
  events/hr | 31.0 (25.0) | 27.2 (24) | 29.1 (24.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Adhering to Positive Airway Pressure (PAP)
Description: PAP adherence will be measured from the PAP unit (which monitors nightly hours of use and records this data; this is the standard of care clinical practice approach used currently by health care providers to monitor PAP use) and will be reported as Number of Participants who Adhered to Positive Airway Pressure (PAP) Treatment (adherence defined as >4 hours of use per night on average across the 30 day period). For example, if 5 subjects used PAP for more than 4 hours per night on average across the 30 day period, then the number of adherent participants is 5.
Time Frame: one month
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Groups:
- Control: Standard Care: Standard care: This is the care that would be routinely provided by their healthcare provider
Arm/Group | Intervention: AirCare System | Control: Standard Care
Number analyzed (Participants) | 74 | 72
Participants | 5 | 3
Statistical Analysis 1: Comparison: Intervention: AirCare System vs Control: Standard Care; Test type: Superiority; p = 0.72, Chi-squared

ADVERSE EVENTS:
Time Frame: One month
Description: Adverse events were collected at the one month follow-up visit
Arm/Group | Intervention: AirCare System | Control: Standard Care
All-Cause Mortality (participants affected / at risk) | 3/74 | 4/72
Serious Adverse Events (participants affected / at risk) | 17/74 | 17/72
Other Adverse Events (participants affected / at risk) | 1/74 | 4/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention: AirCare System (N=74) | Control: Standard Care (N=72)
Aortic Stenosis (Cardiac disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Atrial Fibrillation (Cardiac disorders) | 1 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
CAD (Cardiac disorders) | 4 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Cardiac Arrest (Cardiac disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
CHF (Cardiac disorders) | 13 | 10 — Related? (U=Unrelated, R=Related): U / Expected? Y
Hypotension (Cardiac disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Pacemaker bleeding (Cardiac disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Pacemaker malfunction (Cardiac disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
PVT (Cardiac disorders) | 2 | 2 — Related? (U=Unrelated, R=Related): U / Expected? Y
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Abnormal Liver Enzymes (Gastrointestinal disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
GI Bleed (Gastrointestinal disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Sepsis (Infections and infestations) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
SIRS (Infections and infestations) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
CVA (Nervous system disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Neuropathy (Nervous system disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Seizure (Nervous system disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Stroke (Nervous system disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Syncope (Nervous system disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Kidney infection (Renal and urinary disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention: AirCare System (N=74) | Control: Standard Care (N=72)
Urinary Tract Infection (Infections and infestations) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Diarrhea (Gastrointestinal disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Toothache (General disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Atrial Fibrillation (Cardiac disorders) | 0 | 1 — Related? (U=Unrelated, R=Related): U / Expected? Y
Lightheadedness (Nervous system disorders) | 1 | 0 — Related? (U=Unrelated, R=Related): U / Expected? Y

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT02312765/Prot_SAP_000.pdf